CLINICAL TRIAL: NCT03912051
Title: Assessment of Performance and Safety of an Asymmetric Balloon in the Treatment of Intranasal Bleeding Managed in an Emergency Setting
Acronym: BATSI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Dianosic (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: DEF2018
Record Dates: First submitted 2019-04-08; First posted 2019-04-11 (Actual); Last update posted 2019-09-03 (Actual); Status verified 2019-08

CONDITIONS: Epistaxis
MeSH Terms: conditions — Epistaxis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- asymmetric balloon (Experimental): Asymmetric air filled (max 25 cc, Leur lock syringe) epistaxis balloon
  Interventions: Device: asymmetric balloon

INTERVENTIONS:
Device: asymmetric balloon — Asymmetric balloon for treatment of intranasal bleeding
  Other Names: epistaxis balloon

SUMMARY:
Between 10 and 12% of the general population suffers from epistaxis, out of which 10% would need to be medically managed. Most of patients treated for epistaxis are managed through emergency departments. The involvement of the ENT (ear, nose and throat) surgeon might be required in more complex situations in order to control bleeding.

Usually, nasal packing packing is used as a first line option after failure of digital compression. Epistaxis balloons are often used after failure of nasal packing Balloons are effective in approximately 60% of the patients with a rapid control of bleeding by compression followed by an absence of rebreeding after balloon removal.

The main challenges for patients treated with this device are i) pain upon balloon introduction and inflation ii) discomfort upon introduction in the nasal cavity as well as during balloon maintenance during 24 to 72 hours of tamponade iii) blood retention between distal and proximal balloons that favors infection iv) limited breathing capabilities through the nostrils which increases general discomfort v) negative aesthetic impact for the patient vi) septal and alar necrosis risk in case of prolonged compression.

Moreover, epistaxis leading to an hospitalization between 24 to 48h are not rare (>11 000 in France in 2017 according to ATIH). Those hospitalizations are often decided in order to ensure an optimal patient monitoring following packing or epistaxis balloon placement.

In order to address those adverse events while keeping the same efficacy and avoiding hospitalizations or reducing their duration, the use of an asymmetric, more physiological, easy to use and mainly intranasal (discreet proximal extremity) is studied.

ELIGIBILITY:
Inclusion Criteria:

* Age > or = 18 years
* Male and female
* bleeding uncontrolled with digital compression
* Patient registered at social security
* Patient who gave informed consent

Exclusion Criteria:

* Allergy to xylocaine
* Impossibility to give patient information (severe massive epistaxis, difficulty to understand, non awaken patient…)
* Patient in custody of court
* Patient under guardianship or curator

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2019-03-27 (Actual); Primary Completion 2019-06-30 (Actual); Study Completion 2019-07-18 (Actual)

PRIMARY OUTCOMES:
Device performance | 12 days
  Absence of bleeding following balloon inflation during first 48 hours and absence of rebreeding following removal at 48 hours and 9 days following removal
Device safety | 12 days
  Pain score on a VAS (Visual Analogic Scale)

SECONDARY OUTCOMES:
QoL | 12 days
  RhinoQoL (Rhino Quality of Life) score

CONTACTS AND LOCATIONS:
Overall Officials: Christian Debry, Pr, Principal Investigator — CHU Strasbourg (Univ Hosp Strasbourg)
Locations (1):
- CHU Strasbourg, Strasbourg, Grand Est, France

IPD SHARING:
Plan to Share IPD: No